CLINICAL TRIAL: NCT02594813
Title: Bleeding Rate After EGD and Colonoscopy in Patients Who Continue to Take Antithrombotic Agents
Acronym: EGD
Status: Recruiting | Type: Observational
Sponsor: Showa Inan General Hospital (Other)
Responsible Party: Principal Investigator, Akira Horiuchi, Chief, Showa Inan General Hospital
Other Study IDs: Bleeding rate
Record Dates: First submitted 2015-10-30; First posted 2015-11-03 (Estimated); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Bleeding After GI Endoscopy
MeSH Terms: interventions — Biopsy; Cold Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Excised specimens after taking biopsy or doing polypectomy
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Biopsy, cold or hot snare polypectomy, or EMR

SUMMARY:
The bleeding rate of both EGD (including biopsy) and colonoscopy (including biopsy, cold or hot snare polypectomy, or EMR) in patients who continue to take various antithrombotic drugs is studied prospectively. The immediate or delayed bleeding that requires hemostatic clipping or other endoscopic treatments is defined as the bleeding. Immediate bleeding requiring hemostatic clipping is defined as spurting or oozing which continued for more than 30 seconds. Delayed bleeding is defined as bleeding that requires the endoscopic treatment within 2 weeks after endoscopy. Prophylactic clipping is not performed after taking biopsy and doing polypectomy. Additionally, investigators evaluate the rate of injured submucosal arteries of the excised specimen when the bleeding occurs.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria is all patients who continue to take antithrombotic drugs and undergo EGD or colonoscopy

Exclusion Criteria:

* Patients who take prophylactic clipping after biopsy or polypectomy American Society of Anesthesiologists physical status of class IV or V

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients who continue to take antithrombotic drugs undergo EGD including biopsy and colonoscopy including biopsy, snare or hot polypectomy and/or EMR.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2015-11; Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
the rate of delayed bleeding | 10 years
  Delayed bleeding defined as bleeding that required endoscopic treatment within 2 weeks after the procedure.

SECONDARY OUTCOMES:
the rate of immediate bleeding | 10 years
  Immediate bleeding defined as spurting or oozing which continued for more than 30 seconds.
the number of clip used | 10 years
  The number of clip used during the procedures.

CONTACTS AND LOCATIONS:
Overall Officials: Akira Horiuchi, MD, Principal Investigator — Showa Inan General Hospital
Locations (1):
- Showa Inan General Hospital, Komagane, Japan

REFERENCES:
- [Derived] Nonaka E, Horiuchi I, Horiuchi A, Ukai S, Takahata N, Oishi K. The Risk of Colonoscopy-related Bleeding in Patients With or Without Continued Treatment With an Antithrombotic Agent. DEN Open. 2025 Jul 17;6(1):e70175. doi: 10.1002/deo2.70175. eCollection 2026 Apr. PMID 40677618
- [Derived] Morita A, Horiuchi I, Tanaka N, Takada H, Graham DY, Horiuchi A. Managing bleeding risk after cold snare polypectomy in patients receiving direct-acting oral anticoagulants. Gastrointest Endosc. 2022 May;95(5):969-974. doi: 10.1016/j.gie.2022.01.005. Epub 2022 Jan 19. PMID 35065046